CLINICAL TRIAL: NCT06928753
Title: Real-world Effectiveness, Safety and Immunogenicity of Chikungunya Vaccination in Populations at Risk of Severe or Complicated Forms: Prospective Study in La Réunion
Acronym: CHIK-RE-VAC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government); Région La Réunion (Unknown); ARS La Réunion (Unknown); Direction Générale de l'offre de Soins (DGOS) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025/CHU/12; 2025-521307-43-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-04

CONDITIONS: Chikungunya Virus Infection
Keywords: Prophylaxis, Safety, Efficacy, Vaccine effectiveness, Chikungunya
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaccinated group (Experimental): Patients who will be vaccinated with the IXCHIQ vaccine
  Interventions: Biological: IXCHIQ
- Non-vaccinated group (No Intervention): Patient who will not be vaccinated

INTERVENTIONS:
Biological: IXCHIQ — Group of vaccinated arm will be with the IXCHIQ vaccine
  Arms: Vaccinated group

SUMMARY:
Against the backdrop of a growing chikungunya epidemic in La Réunion, this prospective study will assess the real-life efficacy, safety and immunogenicity of IXCHIQ® vaccine in vulnerable individuals (seniors, comorbid patients), defined by the French Health Autority (HAS) as at risk of severe or complicated forms and/or chronic disabling forms (chronic arthritis, chronic fatigue phenotypes). This study will also provide input for the preparation of a cluster randomized trial on a population scale.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for anti-chikungunya vaccination according to french Health Authority (HAS)
* Beneficiary of social security coverage
* Signature of informed consent form

Exclusion Criteria:

* Pregnant women
* Vaccine contraindication for patients undergoing medical treatment
* Persons under guardianship, curatorship or safeguard of justice
* Anyone who has received immunoglobulin or a blood or plasma transfusion 3 months prior to vaccine administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To measure the vaccine effectiveness at 6 months | 6 months
  Vaccine effectiveness defined at 6 months as the difference in attack rate between unvaccinated and vaccinated participants divided by the attack rate in unvaccinated participants

CONTACTS AND LOCATIONS:
Overall Officials: Patrick GERARDIN, MD, Study Director — CHU La Réunion
Locations (1):
- CHU La Réunion, Saint-Denis, France